CLINICAL TRIAL: NCT06057207
Title: Effects of Perioperative Circulating Adiponectin Levels on Postoperative Systemic Inflammatory Response in Patients Undergoing Major Colorectal Surgery
Brief Title: Perioperative Blood Adiponectin Dynamics and Systemic Infflamatory Response After Major Colorectal Surgery
Acronym: ADIPOS
Status: Completed | Type: Observational
Sponsor: Osijek University Hospital (Other)
Responsible Party: Principal Investigator, Sonja Skiljic, Principal Investigator, Osijek University Hospital
Other Study IDs: ADIPOS study
Record Dates: First submitted 2023-09-19; First posted 2023-09-28 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Obesity, Abdominal; Surgery; Systemic Inflammatory Response Syndrome; Postoperative Complications; Colorectal Carcinoma (CRC); Adiponectin
Keywords: adiponectin; IL-6; obesity; surgery; systemic infflamatory response syndrome; colorectal carcinoma; final outcome
MeSH Terms: conditions — Obesity, Abdominal; Systemic Inflammatory Response Syndrome; Postoperative Complications; Colorectal Neoplasms; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples from every patient will be taken preoperatively, 24 hours and 72 hours postoperatively.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- all patients presenting for elective open colorectal resection due to colorectal carcinoma
  Interventions: Diagnostic Test: serum levels of adiponectin; Diagnostic Test: IL-6; Other: Postoperative systemic infflamation; Other: Postoperative complications

INTERVENTIONS:
Diagnostic Test: serum levels of adiponectin — adiponectin level will be measured on a day of surgery, 24 hours and 72 hours after surgery
Diagnostic Test: IL-6 — IL-6 level will be measured on a day of surgery, 24 hours and 72 hours after surgery
Other: Postoperative systemic infflamation — systemic infflamatory response syndrome (SIRS) will be estimated in firs 72 hours after surgery by clinical criteria: apperance of at least 2 from 4 major clinical signs of SIRS: heart rate>90/min, body temperature >38 C or <36 C, WBC >12 000 or <4000, hyperventilation, CRP >50mg/L, PCT > 0.5 ug/L.
Other: Postoperative complications — Complications in early postoperative period during hospitalisation will be including: surgical operation site related: anastomotic or laparotomic dehiscence, wound/local infection, postoperative bleeding, reoperation and nonsurgical site complications: sepsis, pneumonia, noncardiac respiratory failure, (need for noninvasive oxygen therapy), prolonged mechanical ventilation >24 hours postoperative, reintubation, repeated mechanical ventilation atrial fibrillation, congestive heart failure, myocardial infarction, acute kidney injury/failure, postoperative delirium. Length of ICU and overall hospital stay with after discharge from hospital will be documented.

SUMMARY:
Surgical stress after major abdominal surgery in perioperative period causes neuroendocrine, metabolic and imunologic changes in organism with production of proinfflamatory citokines and results with appearance of systemic infflammmatory response syndrome (SIRS). Dysregulated and overrated SIRS in early postoperative period can lead to complications with additional comorbidities, longer hospital stay and poorer outcome. A low grade chronic infflammatory state in obesity and hypoadiponectinemia can enable the cytokine storm and exaggerated /dysregulated SIRS in obese patients after surgery. Obesity according to this knowledge presents independent risk factor for developing more severe systemic infflamatory response syndrome in early postoperative period after major abdominal surgery. Also, chronic intestinal and gut infflamation is leading theory in oncogenesis of colorectal carcinoma according to recent findings. Many studies find low adiponectin levels in patients with colorectal carcinoma compared to healthy population. Obesity and colorectal cancer have infflamation and low adiponectin level as mutual factor which can be the important key in pathophysiology process of colorectal oncogenesis which are extremly complicated , multifactorial and intertwining.

Hypothesis: Lower blood adiponectin levels are associated with higher systemic infflamatory response in patients after major abdominal surgery. Major aim of this study is to investigate correlation between perioperative blood levels of adiponectin and clinical signs of systemic infflamation and blood markers of systemic infflamation in patients after major colorectal surgery.

DETAILED DESCRIPTION:
Gastrointestinal tumors are commonly presented for surgical resections. According to Global Cancer Statistics 2020: GLOBOCAN estimates colorectal carcinoma ranks third in terms of incidence, but second in terms of mortality for overall carcinomas worldwide. At the same time, obesity is a fast growing disease with of pandemic proportions with a current global prevalence of 39% according to the World Health Organisation (WHO). Many patients presented for major abdominal resections of colrectal carcinomas are obese. Obesity is chronic disease with complex pathophisiology. Adipose tissue besides being a storage site is responsible for secretion of various adipokines with imunometabolic role. Adipokines (also called adipocytokines) are cell-signaling molecules (cytokines) produced by the adipose tissue that play many functional roles in energy/metabolic status of the body, and inflammation. Among adipokines, adiponectin is predominantly antiinfflamatory adipokine which inhibits production of infflammatory citokines (IL-6) and is decreased in obesity. Adipocyte dysfunction in obesity with altered adipokines release results in chronic low-grade inflammatory state. Obesity is also well known risk factor for colorectal carcinoma in which oncogenesis adiponectin may be the important key according to recent findings.

Surgical stress after major colorectal surgery in perioperative period causes neuroendocrine, metabolic and imunologic changes in organism with production of proinfflamatory citokines and results with appearance of systemic infflammmatory response syndrome (SIRS). Dysregulated and overrated SIRS in early postoperative period can lead to complications with additional comorbidities, longer hospital stay and poorer outcome. A low grade chronic infflammatory state in obesity and colorectal carcinoma associated with potential hypoadiponectinemia can enable the cytokine storm and exaggerated /dysregulated SIRS in these patients after surgery. Due to this knowledge, it is logical to presume that adiponectin levels in perioperative period are associated with the intensity of systemic infflamatory response after major colorectal surgery.

Hypothesis: Perioperative blood adiponectin levels are associated with higher intensity of systemic infflamatory response in patients after major colorectal surgery.

Aim of this study is to:

1. Measure and investigate correlation between perioperative blood adiponectin levels and appearance and intensity of systemic infflamatory response in patients after major colorectal surgery.
2. Investigate correlation between perioperative blood adiponectin levels, SIRS and postoperative complications, days of ICU and lenght of hospital stay in patients presenting for major colrectal surgery.

Research plan: After ethical approval and written informed consent, demographic, antropometric and comorbidities data will be taken from all patients included in study. BMI, waist circumference and ultrasound measurments of abdominal fat thickness ( superficial and visceral abdominal fat thickness) will be taken preoperatively. Blood collections for determining adiponectin levels, IL-6, Complete Blood Count with Differential Blood Count, lactats in arterial blood, C-reactive protein(CRP), procalcitonin(PCT), albumins (ALB), neutrophil/lymphocite ratio (NLR), platelet/lymphocyte ratio (PLR), CRP/ALB ratio, Systemic Immune-Inflammation Index (SII), Systemic inflammation response index (SIRI) will be taken before surgery (1), 24 hours after surgery (2) and 72 hours after surgery (3). All patients will bi given the same technique of balanced general endotracheal anesthesia with the same drugs and the same postoperative multimodal analgesia regimen. Appearance of SIRS in first 72 hours postoperative period will be detected and documented according to standardized major clinical SIRS criteria. Complications in early postoperative period during hospitalisation will be including: surgical operation site related according to standardized Clavien-Dindo classification: anastomotic dehiscence, wound/local infection, postoperative bleeding, reoperation and systemic complications: sepsis, pneumonia, noncardiac respiratory failure, (need for noninvasive oxygen therapy), prolonged mechanical ventilation >24 hours postoperative, reintubation, repeated mechanical ventilation, cardiovascular complications: atrial fibrillation, congestive heart failure, myocardial infarction, acute kidney injury/failure, postoperative delirium presence. After surgery, histological tumor grade, pathohistological tumor staging ( 8th edition of the American Joint Committee on Cancer (AJCC) staging) and tumor localisation ( colon/rectum) will be documented.

Length of ICU and overall hospital stay with outcome of surviving or death after discharge from hospital will be documented.

Significance/Expected scientific contribution: Understanding of the underlying pathophysiological mechanisms which contributes to the appearance and severity of SIRS with possible complications in early postoperative period is important for developing more predictive diagnostics and possible treatment options for improvements in outcome especially in major surgical procedures. The adipocytokines have important role in many aspects of inflammation and immunity. This study can help in better understanding the infflamatory role od adiponectin in pathophysiology of SIRS after major colorectal surgery.

ELIGIBILITY:
Inclusion Criteria:

Diagnose of colorectal cancer Age >18 years Patient presenting for major (open) elective colorectal surgery according to carcinoma.

Written informed consent.

Exclusion Criteria:

Age<18 years BMI<18.5kg/m2 Acute surgical conditions Established acute systemic/local infection Chronic/actual corticosteroid therapy Active immunomodulation therapy Allergie to used anestehetics/analgetics in study. Patient refusal Laparoscopic surgery Massive intraoperative surgical bleeding Preexisting concomitant second carcinoma other than colorectal origin Patients which does not fulfill inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting for major (open) elective colorectal surgery of colorectal carcinoma
Sampling Method: Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2023-07-27 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-08-22 (Actual)

PRIMARY OUTCOMES:
Adiponectin | Preoperative, 24 hours after surgery, 72 hours after surgery
  Three measurements of adiponectin will be taken from blood samples of every patient preoperative, 24 and 72 hours postoperative

SECONDARY OUTCOMES:
IL-6 | Preoperative, 24 hours after surgery, 72 hours after surgery
  Three measurements of IL-6 will be taken from blood samples of every patient preoperative, 24 and 72 hours postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Slavica Kvolik, Study Director — Department of Anaesthesiology, Resuscitation and ICU, Osijek University Hospital,
Locations (2):
- Croatia (2):
  - Osijek University Hospital, Osijek, Osijek
  - Sonja Škiljić, Osijek, Osijek

IPD SHARING:
Plan to Share IPD: Undecided
After study completion, upon reasonable request, data may be shared with other researchers.

REFERENCES:
- [Background] Florescu A, Branisteanu D, Bilha S, Scripcariu D, Florescu I, Scripcariu V, Dimofte G, Grigoras I. Leptin and adiponectin dynamics at patients with rectal neoplasm - Gender differences. PLoS One. 2019 Aug 19;14(8):e0212471. doi: 10.1371/journal.pone.0212471. eCollection 2019. PMID 31425509
- [Background] Boersema GSA, Wu Z, Menon AG, Kleinrensink GJ, Jeekel J, Lange JF. Systemic Inflammatory Cytokines Predict the Infectious Complications but Not Prolonged Postoperative Ileus after Colorectal Surgery. Mediators Inflamm. 2018 Mar 6;2018:7141342. doi: 10.1155/2018/7141342. eCollection 2018. PMID 29692682
- [Background] Barbic J, Ivic D, Alkhamis T, Drenjancevic D, Ivic J, Harsanji-Drenjancevic I, Turina I, Vcev A. Kinetics of changes in serum concentrations of procalcitonin, interleukin-6, and C- reactive protein after elective abdominal surgery. Can it be used to detect postoperative complications? Coll Antropol. 2013 Mar;37(1):195-201. PMID 23697273
- [Background] Neskovic N, Mandic D, Marczi S, Skiljic S, Kristek G, Vinkovic H, Mraovic B, Debeljak Z, Kvolik S. Different Pharmacokinetics of Tramadol, O-Demethyltramadol and N-Demethyltramadol in Postoperative Surgical Patients From Those Observed in Medical Patients. Front Pharmacol. 2021 Apr 15;12:656748. doi: 10.3389/fphar.2021.656748. eCollection 2021. PMID 33935773
- [Background] Wei Y, Zhu F, Gong J, Yang J, Zhang T, Gu L, Zhu W, Guo Z, Li Y, Li N, Li J. High Visceral to Subcutaneous Fat Ratio Is Associated with Increased Postoperative Inflammatory Response after Colorectal Resection in Inflammatory Bowel Disease. Gastroenterol Res Pract. 2018 Apr 3;2018:6270514. doi: 10.1155/2018/6270514. eCollection 2018. PMID 29849595
- See also: Leptin and adiponectin dynamics at patients with rectal neoplasm - Gender differences. — https://pubmed.ncbi.nlm.nih.gov/31425509/
- See also: Systemic Inflammatory Cytokines Predict the Infectious Complications but Not Prolonged Postoperative Ileus after Colorectal Surgery. — https://pubmed.ncbi.nlm.nih.gov/29692682/
- See also: Kinetics of changes in serum concentrations of procalcitonin, interleukin-6, and C- reactive protein after elective abdominal surgery. Can it be used to detect postoperative complications? — https://pubmed.ncbi.nlm.nih.gov/23697273/
- See also: Different Pharmacokinetics of Tramadol, O-Demethyltramadol and N-Demethyltramadol in Postoperative Surgical Patients From Those Observed in Medical Patients. — https://pubmed.ncbi.nlm.nih.gov/33935773/
- See also: High Visceral to Subcutaneous Fat Ratio Is Associated with Increased Postoperative Inflammatory Response after Colorectal Resection in Inflammatory Bowel Disease — https://pubmed.ncbi.nlm.nih.gov/29849595/